CLINICAL TRIAL: NCT02352025
Title: A Pre-surgical Clinical Trial of Therapy With S-equol in Women With Triple Negative Breast Cancer.
Brief Title: S-equol in Women With Triple Negative Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 14-2018; HSC20150231H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: S-equol; breast cancer; triple negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Equol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-equol (Experimental): After having a core needle biopsy of the breast confirming triple negative breast cancer, eligible women enrolled on the study will be treated with S-equol at a dose of 50 mg PO twice daily for 14 days.
  Interventions: Drug: S-equol

INTERVENTIONS:
Drug: S-equol — S-equol should be administered orally, twice daily (12 hours apart), preferably on an empty stomach with a glass of water. Tablets should be swallowed whole.
  Other Names: Equol

SUMMARY:
The primary objective of this study is to determine if S-equol, an ER-beta agonist, is effective in decreasing the proliferation rate of triple negative breast cancer.

DETAILED DESCRIPTION:
After a baseline breast tumor core biopsy, eligible women with triple negative breast cancer (ER- alpha, PR and HER-2 receptor negative) will be treated with S-equol at a dose of 50 mg twice daily for a period of about 14 days (10-21 day range). After completion of treatment, a second breast tumor sample will be obtained to compare molecular changes between the two specimens. The second pathology specimen may be from the surgical resection of the breast tumor, or a repeat core needle biopsy, if no further surgery is planned. The primary endpoint will be the absolute change in the Ki67, which is a validated marker of tumor proliferation in breast cancer. Secondary endpoints will include assessment of total ER-beta and pY36 levels as measured by immunohistochemical staining and their correlation with S-equol effects. Further treatment after surgical resection or second core needle biopsy of the tumor will be guided by tumor size, nodal status and other standard parameters, and is at the discretion of the treating physician. The Investigator hypothesizes that S-equol will cause a measurable decrease in Ki-67 in estrogen receptor beta expressing triple negative breast cancers, indicating its potential efficacy in this tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be women who are 18 years old or older.
* Ability to consent to treatment - patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* Previously untreated breast cancer determined by a core needle biopsy showing invasive ductal carcinoma or invasive lobular carcinoma.
* A prior, unrelated, breast cancer is allowed.
* All stages of breast cancer are eligible.
* Estrogen receptor negative - defined as less than or equal to 5% staining by IHC.
* Progesterone receptor negative - defined as less than or equal to 5% staining by IHC.
* HER 2 negative as defined as 2+ or less using IHC or a ratio of less than 2.0 on FISH testing.
* Patient must be able to take oral medications. Patients may not have any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study drug.
* Patients may not be pregnant or breast feeding.
* Patients must with eligible for surgical resection of their breast cancer or repeat biopsy after completing 14 days of treatment.
* Patients must have a complete history and physical examination within 28 days prior to registration.
* Patients must have a performance status of ECOG 0, 1, 2.
* Patient may not be concurrently enrolled in another investigational drug treatment study.
* Tissue block of initial biopsy specimen is available.

Exclusion Criteria:

* Known hypersensitivity to S-equol or any of its excipients.
* ECOG status 3 or 4.
* As judged by the investigator, severe uncontrolled concurrent medical conditions, psychiatric illness or social condition that would limit compliance with study requirements.
* Evidence of any significant clinical disorder or laboratory finding that makes it undesirable for the subject to participant in the clinical trial.
* Any prior treatment for the current, newly diagnosed breast cancer.
* Current use of SERMS or aromatase inhibitors.
* Inflammatory breast cancer or patients with rapidly progressing metastatic breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Proliferation Rate of Triple Negative Breast Cancer | 14 Days
  Biopsy will measured by change in Ki-67

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lathrop, MD, Principal Investigator — principle investigator
Locations (1):
- CTRC (Cancer Therapy and Research Center) at UTHSCSA, San Antonio, Texas, United States